CLINICAL TRIAL: NCT05343884
Title: NUCLEuS: Evaluating DyNamic Myocardial Blood Flow QUantitation As a Cost Effective Care ModeL for DiabEtic Patients With Coronary Artery DiSease: A Randomized Controlled Trial
Brief Title: Evaluating DyNamic Myocardial Blood Flow QUantitation As a Cost Effective Care ModeL for DiabEtic Patients With Coronary Artery DiSease
Acronym: NUCLEuS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart Centre Singapore (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021/2780
Record Dates: First submitted 2022-03-15; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Coronary Artery Disease; Diabetes Mellitus
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dynamic myocardial perfusion imaging (Other): Dynamic myocardial perfusion imaging is performed to obtain additional measurements of coronary blood flow, compared to conventional imaging.
  Interventions: Radiation: Myocardial perfusion imaging
- Conventional myocardial perfusion imaging (Other): Conventional myocardial perfusion imaging which is based on standard routine clinical myocardial perfusion imaging.
  Interventions: Radiation: Myocardial perfusion imaging

INTERVENTIONS:
Radiation: Myocardial perfusion imaging — Myocardial perfusion imaging

SUMMARY:
This will be a prospective randomized clinical trial comprising of n=300 diabetic patients, randomized to either dynamic (n=150) or conventional MPI (n=150) strategy. Healthcare resources utilization of each patient will be tracked. Patients will be followed up for short term outcomes and for long term outcomes.

DETAILED DESCRIPTION:
Diabetes mellitus poses unique problems to detection and management of coronary atherosclerosis. Among the diabetics, certain spectrums of coronary atherosclerosis may be missed on conventional myocardial perfusion imaging, such as early coronary microvascular dysfunction. On the other spectrum, advanced coronary atherosclerosis may result in balanced ischemia, recording falsely negative results on conventional myocardial perfusion imaging. These uncertainties either lead to more downstream testing or under-detection resulting in higher risks of adverse outcomes. Compared to conventional myocardial perfusion imaging (MPI), dynamic MPI quantitation is a new validated technique that provides additional quantitation across the entire spectrum of coronary atherosclerosis.

Outcomes:

Short term outcomes:

* The primary end-point is diagnostic failure, defined as unnecessary coronary angiography (absence of ≥50% stenosis in ≥1 coronary arteries) or any additional coronary testing (example, computed tomography of coronary arteries).
* Secondary end-points are post-test referral to coronary angiography, coronary revascularization (percutaneous coronary intervention or coronary artery bypass surgery), or escalation in anti-anginal medication.

Long term outcomes:

* Major adverse cardiovascular events to be measured include cardiac mortality, acute myocardial infarction, unstable angina, any revascularization, up till 36 months.
* Quality of life (QOL): Using Seattle Angina Questionnaire (SAQ) and EuroQOL-5D-3L, we will measure the difference in QOL measured at baseline and follow-up within each diagnostic strategy, and compared between both strategies.

The differences in healthcare resource utilization and associated costs will be compared between the two diagnostic strategies.

Group A

Visit 1 and/or Visit 2:

Baseline procedures

1. Cardiovascular measurements:

   Non-invasive brachial blood pressure machine Echocardiogram Standard transthoracic echocardiographic examination will be performed according to established laboratory practice using standard commercially available machines.

   Resting electrocardiography will be performed to ascertain sinus rhythm.
2. Biospecimen collection Fresh blood, urine and/or stool specimens will be collected for biochemistry, biomarkers and other profiles.
3. Musculoskeletal and Physical Analysis Participants will undergo focused examinations that include measurement of height, weight, body mass index, waist circumference, body composition analysis and handgrip strength.
4. Questionnaires You will be interviewed by our study coordinator regarding your health condition and other questions related to your health, physical activity and lifestyle and other questionnaires.
5. Dynamic myocardial perfusion imaging Dynamic myocardial perfusion imaging is performed to obtain additional measurements of coronary blood flow, compared to conventional imaging.

Group B

Visit 1 and/or Visit 2:

Baseline procedures

1. Cardiovascular measurements:

   Non-invasive brachial blood pressure machine Echocardiogram Standard transthoracic echocardiographic examination will be performed according to established laboratory practice using standard commercially available machines.

   Resting electrocardiography will be performed to ascertain sinus rhythm.
2. Biospecimen collection Fresh blood, urine and/or stool specimens will be collected for biochemistry, biomarkers and other profiles.
3. Musculoskeletal and Physical Analysis Participants will undergo focused examinations that include measurement of height, weight, body mass index, waist circumference, body composition analysis and handgrip strength.
4. Questionnaires You will be interviewed by our study coordinator regarding your health condition and other questions related to your health, physical activity and lifestyle and other questionnaires.
5. Conventional myocardial perfusion imaging You will undergo conventional myocardial perfusion imaging which is based on standard routine clinical myocardial perfusion imaging.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients without known coronary artery disease referred for MPI

Exclusion Criteria:

* History of percutaneous coronary intervention, coronary artery bypass graft surgery
* Asthma
* Chronic obstructive pulmonary disease (COPD)
* Presence of cardiac devices such as pacemakers and implantable cardiac defibrillators

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Failure | Up to 12 months
  The primary end-point is diagnostic failure, defined as unnecessary coronary angiography (absence of ≥50% stenosis in ≥1 coronary arteries) or any additional coronary testing (example, computed tomography of coronary arteries).

SECONDARY OUTCOMES:
Secondary end-points | Up to 12 months
  Secondary end-points are post-test referral to coronary angiography, coronary revascularization (percutaneous coronary intervention or coronary artery bypass surgery), or escalation in anti-anginal medication.

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart Centre Singapore, Singapore, Singapore